CLINICAL TRIAL: NCT05083819
Title: Microbiological Assessment of Air and Surfaces of Operation Rooms in Assuit University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Hussien Mahran Shehata, Principal Investigator, Assiut University
Other Study IDs: Microbiological assessment
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Air, Surfaces

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To determine the bacteriological load on air and surfaces within the ORs.
2. To isolate and identify pathogenic strains of bacteria on equipments and contact surfaces.
3. To compare between adenosine triphosphate bioluminescence assay and the ordinary cultures in order to verify whether the methods of hygienization and disinfection implemented were in fact effective.

DETAILED DESCRIPTION:
Healthcare-associated infections often have multiple etiologies, of which cleanliness of hospital surfaces can play a large role. This is perhaps most important in the operating room, where a sterile environment is paramount to decreasing the burden of hospital-acquired morbidity and surgical site infections. Contaminated hospital surfaces greatly contribute to the transmission of healthcare associated pathogens, including methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant Enterococcus spp (VRE), and Clostridium difficile Surgical site infections (SSIs) are infections that occur after surgery in the part of the body where the surgery took place and account for about 14-20% of all hospital-acquired (nosocomial) infections. Some are superficial, involving only the skin, while others are more serious and can involve tissues under the skin, organs, or implanted material. Factors causing SSIs are known to be multifarious. Superficial SSIs are most often associated with environmental factors, such as environmental contamination by fungi and bacteria, surface contamination, humidity, differential pressure and temperature of the OR, while factors that determine deep and organ/space SSIs are more often associated with patient characteristics (age, sex, transfusion, nasogastric feeding and nutrition, as measured by the level of albumin in the blood), type of intervention and preoperative stay .

SSIs continue to be a major problem in modern medicine, with both individual and economic consequences. They are the most frequent nosocomial infections in low- and middle-income countries, affecting up to one third of patients who have undergone a surgical procedure, while in high-income countries they are the second most frequent type .

Contaminated surfaces and fomites are considered an important reservoir of (multi-resistant) microorganisms in hospitals. Therefore, cleaning of the environment is important for reducing bacterial spread, controlling antimicrobial resistance and improving patient .

Air quality in ORs should be assessed during microbiological commissioning of new ORs and whenever required thereafter. OR ventilations are very much variable from country to country, within a country and even within a hospital as per requirement and availability. Ventilation systems are classified as conventional plenum ventilation (CV), laminar flow ventilation (LAF), wall mounted air conditioners and free-standing air conditioners.

Microbial monitoring of ORs (and also of other controlled environments, such as recovery rooms) is therefore essential to obtain representative estimates of the bioburden of the environment. It includes quantitation of the microbial content of room air, compressor air that enters the critical area, surfaces, equipment, sanitization containers, floors, walls and personnel garments and also the search for Legionella pneumophila in the water systems. Information gathered from the data compiled and analysed can then be useful in the investigation of the source of the contamination and the subsequent adoption of preventive measures.

The assessment of the cleanliness of surfaces in hospitals is mostly conducted by visual inspection. This method is not sensitive and subjective and therefore unreliable. Recently, a more objective technique was introduced to measure biological contamination. This technique is based on the measurement of adenosine triphosphate (ATP), a molecule that is present in all organic cells.

Traditional microbiological techniques are the most commonly used methods to evaluate hygienic quality, but they require specific skills, long execution and analysis times and are therefore unsuitable for routine monitoring. In the last decade alternative methods for assessing environmental cleanliness have been proposed, including the adenosine triphosphate (ATP) bioluminescence assay,based on the measurement of levels of ATP present on an environmental surface. Bioluminescence test exploits the chemiluminescence properties of luciferin-luciferase reagent, which reacts with any ATP residue present on a substrate, emitting light and measuring the presence of organic matter.

The air Sampler is a high-performance instrument that is based on the principle of the Andersen air sampler, which aspirates air through a perforated plate. The resulting airflow is directed onto a 90 mm Petri dish containing agar. For each air sample collection, the air Sampler equipment is placed on a firm support at about 1 m above the ground, the perforated lid is opened by rotating to the right and cleaned with isopropanol. Next, a closed 90 mm Petri dish filled with agar isplaced on top of the dish support, the lid was taken off the Petri dish, the air Sampler perforated lid is closed, the angle of the sampling head is adjusted and the equipment is programmed to aspire 500 L of air (flow rate of 100L/min). After the collection cycle, the sampling head is opened and the Petri dish is closed with the Petri dish cover and placed in the cooler to later be transported to the laboratory.

Microbial monitoring of ORs (and also of other controlled environments, such as recovery rooms) is therefore essential to obtain representative estimates of the bioburden of the environment. It includes quantitation of the microbial content of room air, compressor air that enters the critical area, surfaces, equipment, sanitization containers, floors, walls and personnel garments and also the search for Legionella pneumophila in the water systems. Information gathered from the data compiled and analysed can then be useful in the investigation of the source of the contamination and the subsequent adoption of preventive measures.

Since then research has provided evidence of the importance of establishing environmental monitoring programs to control and maintain an aseptic hospital environment, especially in operating rooms.

ELIGIBILITY:
Inclusion Criteria:

* The study will be carried out in the operation rooms.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Because there is no patient in our study , the study will be carried out on these samples which classified into the following groups as follows:
  * Group 1: 100 samples before starting the surgery in the morning
  * Group 2: 100 samples between the surgeries **These samples will be taken by ordinary swabs, the adenosine triphosphate bioluminescence and the air sampler.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
1.To determine the bacteriological load on air and surfaces within the ORs. | Baseline
  To isolate and identify pathogenic strains of bacteria on equipments and contact surfaces.

REFERENCES:
- [Background] ALFONSO-SANCHEZ, J. L., MARTINEZ, I. M., MARTíN-MORENO, J. M., GONZáLEZ, R. S. & BOTíA, F. 2017. Analyzing the risk factors influencing surgical site infections: the site of environmental factors. Canadian Journal of Surgery, 60, 155. ALMEIDA, B. I. M. 2017. Microbiological assessment of air and surfaces of surgery rooms from a lisbon hospital. DANCER, S. J. 2008. Importance of the environment in meticillin-resistant Staphylococcus aureus acquisition: the case for hospital cleaning. The Lancet infectious diseases, 8, 101-113. MORA, M., MAHNERT, A., KOSKINEN, K., PAUSAN, M. R., OBERAUNER-WAPPIS, L., KRAUSE, R., PERRAS, A. K., GORKIEWICZ, G., BERG, G. & MOISSL-EICHINGER, C. 2016. Microorganisms in confined habitats: microbial monitoring and control of intensive care units, operating rooms, cleanrooms and the International Space Station. Frontiers in microbiology, 7, 1573. ORGANIZATION, W. H. 2016. Global guidelines for the prevention of surgical site infection, World Health Organization. RICHARD, R. D. & BOWEN, T. R. 2017. What orthopaedic operating room surfaces are contaminated with bioburden? A study using the ATP bioluminescence assay. Clinical Orthopaedics and Related Research®, 475, 1819-1824. SANNA, T., DALLOLIO, L., RAGGI, A., MAZZETTI, M., LORUSSO, G., ZANNI, A., FARRUGGIA, P. & LEONI, E. 2018. ATP bioluminescence assay for evaluating cleaning practices in operating theatres: applicability and limitations. BMC infectious diseases, 18, 1-7. TSHOKEY, T., SOMARATNE, P. & AGAMPODI, S. B. 2016. Comparison of two air sampling methods to monitor operating room air quality and assessment of air quality in two operating rooms with different ventilation systems in the national hospital of Sri Lanka. VAN ARKEL, A., WILLEMSEN, I., KILSDONK-BODE, L., VLAMINGS-WAGENAARS, S., VAN OUDHEUSDEN, A., WAEGEMAEKER, P. D., LEROUX-ROELS, I., VERELST, M., MAAS, E. & VAN OOSTEN, A. 2020. ATP measurement as an objective method to measure environmental contamination in 9 hospitals in the Dutch/Belgian border area. Antimicrobial Resistance & Infection Control, 9, 1-8. VANDINI, A., TEMMERMAN, R., FRABETTI, A., CASELLI, E., ANTONIOLI, P., BALBONI, P. G., PLATANO, D., BRANCHINI, A. & MAZZACANE, S. 2014. Hard surface biocontrol in hospitals using microbial-based cleaning products. PLoS One, 9, e108598. WEBER, D. J., ANDERSON, D. & RUTALA, W. A. 2013. The role of the surface environment in healthcare-associated infections. Current opinion in infectious diseases, 26, 338-344.